CLINICAL TRIAL: NCT07046507
Title: Developing a Handheld Anterior Segment Optical Coherence Tomography Device to Assess Kayser Fleischer Rings in Wilson's Disease
Brief Title: The Exploratory Handheld Optical Coherence Tomography Study in Wilson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Aftab Ala, Principal Investigator, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 333382
Record Dates: First submitted 2025-05-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Wilson Disease
Keywords: kayser fleischer rings
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Intervention Model Description: Non-inferiority exploratory study
Who Masked: Outcomes Assessor
Masking Description: Assessors blinded to patient groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of a fixed anterior segment OCT device to detect Kayser Fleischer ring (Active Comparator)
  Interventions: Diagnostic Test: Diagnostic procedures
- Use of a handheld anterior segment OCT device to detect Kayser Fleischer rings (Active Comparator)
  Interventions: Diagnostic Test: Diagnostic procedures

INTERVENTIONS:
Diagnostic Test: Diagnostic procedures — Diagnostic ability of optical coherence tomography in kayser fleischer rings

SUMMARY:
This is an exploratory study using anterior segment optical coherence tomography (OCT) devices to measure copper in the eye. The investigators hope to use this to diagnosis kayser flesicher rings, an important diagnostic criteria in Wilson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Wilson patients with Kayser Fleischer rings on slit lamp examination and 5 patients without Kayser Fleischer rings on slit lamp examination

Exclusion Criteria:

* Those who do not have a confirmed diagnosis of Wilson's disease and no previous formal slit lamp examination will be excluded from recruitment.
* The investigators will also exclude those patients with known corneal disease, history of intraocular disease, haematological disease, pregnancy, and use of topical or intraocular medication.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | Baseline examination
  Can handheld anterior segment optical coherence tomography (OCT) imaging be used as a reliable and practical methodology in the diagnosis/detection of kayser fleischer rings (KFR) in a non-inferior way compared with slit lamp examination and fixed optical coherence tomography. KFR can be visualised on OCT images in a similar way as they are seem on slit lamp examination.

SECONDARY OUTCOMES:
Measurement of the amount of copper in the eye | Baseline examination
  Using OCT images, can we determine an objective value for the amount of copper present in the eye. There are no current methods to determine this value as this is exploratory work.
Is a handheld OCT device non inferior to a fixed OCT device | Baseline examination
  The investigators will compare whether a handheld OCT device can produce images which are non inferior to a fixed OCT device and able to show the presence of Kayser Fleischer rings.
Can this test detect Kayser Fleischer rings before current standard of care testing | Baseline examination
  Slit lamp examination is the current accepted test for detecting Kayser Fleischer rings in the eye. This can be a subjective examination dependent on operator ability. The investigators will assess whether OCT images can detect Kayser Fleischer rings before they are visible on a slit lamp examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey Country Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not appropriate